CLINICAL TRIAL: NCT01755676
Title: A Prospective Study, Parallel, Double-blind, Multicenter for Evaluation of Efficacy of Orlistat 60 mg as Adjuvant Treatment of Obesity in Adults
Brief Title: Evaluation of Orlistat as Adjuvant Treatment of Obesity in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL60EMS0511
Record Dates: First submitted 2012-12-17; First posted 2012-12-24 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orlistat 60 mg (Experimental)
  Interventions: Drug: Orlistat 60 mg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Orlistat 60 mg — 1 tablet 3 times a day
  Arms: Orlistat 60 mg
Other: Placebo — 1 tablet 3 times a day
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of orlistat 60 mg as adjuvant treatment of Obesity in adults.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent;
* Adults Male and Female ≥ 18 years old;
* Obesity (BMI ≥ 30kg/m2 or ≥ 27 Kg/m2 with associate risk);

Exclusion Criteria:

* Pregnancy and Lactation or women without effective contraception;
* Relevant clinical diseases;
* Obesity associated to genetic syndrome;
* Decompensated Diabetes;
* Psychiatric disorders;
* Alimentary disorders;
* Use of: anorectics, herbal weight loss and/or constipation and laxatives, in the past 30 days;
* Patients using cyclosporine or amiodarone;
* Patients with bowel disease;
* Prior bariatric surgery;
* Anemia;
* Hemoglobinopathies and coagulopathy;
* History of cancer in the past five years;
* Use of corticosteroids, oral or injectable, in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of Orlistat 60 mg associated with diet and exercise in relation to placebo associated with diet and exercise in obesity treatment based on weight loss. | 112 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 112 days

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (5):
  - Centro de Medicina Reprodutiva Dr Carlos Isaia Filho, Porto Alegre, Rio Grande do Sul
  - Loema, Campinas, São Paulo
  - Allergisa, Campinas, São Paulo
  - CIPMED, Jaú, São Paulo
  - Marcio Antonio Pereira Clinica de Endocrinologia, São José dos Campos, São Paulo